CLINICAL TRIAL: NCT04668677
Title: Return to Work and Functional Results of French Soldiers After Anterior Cruciate Ligament Reconstruction
Status: Completed | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PPRC10; 2020-A02234-35 (Other: IDRCB)
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: On-line questionnaire — On-line questionnaire about working life, medical care, functional recovery, quality of life and psychological state.

SUMMARY:
The return to work in the military population after surgical reconstruction of the anterior cruciate ligament (ACL) has been poorly investigated within the French armed forces. Only American studies are available and show that this surgery has a significant impact on the operational capacity of soldiers.

ACL rupture is extremely frequent in active populations. This pathology has already been extensively explored in at-risk populations, particularly in sports. Most studies show that the resumption of sport is greatly affected by this pathology.

Furthermore, an over-risk (10 times greater incidence of ACL rupture) in the military has been demonstrated.

ELIGIBILITY:
Inclusion Criteria:

* Military personnel who underwent first-line ACL reconstruction surgery between January 2014 and May 2019

Exclusion Criteria:

* People who have had ACL reconstruction surgery after initial failure
* People with a multiligamentous knee condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of military personnel who underwent first-line ACL reconstruction surgery in a military hospital (military training hospital Bégin or military training hospital Percy) between January 2014 and May 2019.
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2021-01-06 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who regained their professional competence one year after anterior cruciate ligament (ACL) reconstruction surgery. | 1 year after anterior cruciate ligament (ACL) reconstruction surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital d'Instruction des Armées Percy, Clamart, France

IPD SHARING:
Plan to Share IPD: Undecided